CLINICAL TRIAL: NCT02648620
Title: A Prospective, Multi-Center, Single-Arm Trial to Assess the Safety and Feasibility of the SurModics Drug Coated Balloon in the Treatment of Subjects With De Novo Lesions of the Femoropopliteal Artery
Brief Title: Safety and Feasibility of SurModics SurVeil (TM) Drug Coated Balloon
Acronym: PREVEIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUR15-001
Record Dates: First submitted 2015-12-18; First posted 2016-01-07 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases
Keywords: Paclitaxel; Percutaneous Transluminal Angioplasty; PAD; Peripheral Artery Disease; Pharmacokinetics
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SurVeil Drug Coated Balloon catheter (Experimental): Paclitaxel Coated Balloon catheter for angioplasty
  Interventions: Device: SurVeil Drug Coated Balloon; Procedure: Angioplasty

INTERVENTIONS:
Device: SurVeil Drug Coated Balloon — Angioplasty procedure with the SurModics SurVeil Paclitaxel-Coated, Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter (Paclitaxel-coated PTA Catheter)
  Other Names: SurModics SurVeil
Procedure: Angioplasty — Angioplasty procedure with the SurModics SurVeil Paclitaxel-Coated, Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter (Paclitaxel-coated PTA Catheter)
  Other Names: SurModics SurVeil

SUMMARY:
PREVEIL is a prospective, multi-center, single-arm clinical trial to assess the safety and functionality of the SurModics drug coated balloon (DCB) in the treatment of subjects with symptomatic peripheral artery disease (PAD) due to de novo stenoses of the femoral and popliteal arteries. The trial will enroll up to 15 subjects.

DETAILED DESCRIPTION:
PREVEIL will enroll patients presenting with angiographic evidence of significant stenosis in the femoral or popliteal arteries. All enrolled subjects will be treated with the SurVeil DCB.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to participate in the trial:

* Subject is ≥ 18 years.
* Subject has lifestyle-limiting claudication or rest pain with Rutherford classification 2, 3 or 4.
* Subject has provided written informed consent.
* Subject is willing to comply with study follow-up requirements.
* A de novo target lesion in the femoral or popliteal arteries.
* Target lesion must have angiographic evidence of ≥ 50% stenosis by operator visual estimate.
* Target lesion must be ≤ 90 mm in length (one long lesion or multiple serial lesions) by operator visual estimate. Note: Multiple serial lesions are allowed provided that they can be treated as a single lesion with one balloon.
* Target vessel must have an reference vessel diameter (RVD) of 4 mm to 6 mm by operator visual estimate.
* After pre-dilatation, the target lesion is ≤ 70% residual stenosis, absence of a flow limiting dissection and treatable with a single balloon (lesion length ≤90 mm, limited to 100-mm balloon in EFS).
* A patent inflow artery free from significant stenosis (≥ 50% stenosis) as confirmed by angiography.
* At least one patent native outflow artery to the ankle or foot, free from significant stenosis (≥ 50% stenosis) as confirmed by angiography.

Exclusion Criteria:

Subjects will be excluded from the trial if any of the following criteria are met:

* Subject has acute limb ischemia.
* Subject has Rutherford classification of 0, 1, 5 or 6.
* Subject previously underwent any lower extremity percutaneous transluminal angioplasty (PTA) using a DCB within 3 months.
* Subject has had prior vascular intervention within 2 weeks before the planned study index procedure or subject has planned vascular intervention within 30 days after the study index procedure.
* Subject is pregnant and/or breast-feeding or intends to become pregnant during the time of the study OR subject is a male intending to father children within 60 days of index procedure.
* Life expectancy less than 2 years.
* Subject has a known allergy to contrast medium that cannot be adequately pre-medicated.
* Subject is allergic to ALL antiplatelet treatments.
* Subject has impaired renal function (i.e. serum creatinine level ≥ 2.5 mg/dl).
* Subject is dialysis dependent.
* Subject is receiving immunosuppressant therapy.
* Subject has known or suspected active infection at the time of the index procedure.
* Subject has platelet count < 100,000/mm3 or > 700,000/mm3.
* Subject has white blood cell (WBC) count < 3,000/mm3.
* Subject has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the index procedure.
* Subject is diagnosed with coagulopathy that precludes treatment with systemic anticoagulation and/or dual antiplatelet therapy (DAPT).
* Subject is unable to tolerate blood transfusions because of religious beliefs or other reasons.
* Subject is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.
* Subject is known to be incarcerated, mentally incompetent and/or an alcohol or drug abuser.
* Subject is participating in another investigational drug or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints from this study, or subject is planning to participate in such studies prior to the completion of this study.
* Subject has had major surgical or interventional procedures unrelated to this study within 30 days prior to this study or has planned surgical or interventional procedures within 30 days of entry into this study.
* Previous intervention at the lesion site including previous stenting within 3 cm of the target lesion or previous bypass surgery of the target lesion.
* Previous treatment of the target vessel with thrombolysis or surgery.
* Severe concentric calcification of the target lesion.
* Target lesion involves an aneurysm or is adjacent to an aneurysm.
* Target lesion requires treatment with alternative therapy such as stenting, laser, atherectomy, cryoplasty, brachytherapy or re-entry devices.
* Significant vessel tortuosity or other parameters prohibiting access to the target lesion.
* Presence of thrombus in the target vessel.
* Iliac inflow disease requiring treatment , unless the iliac artery disease is successfully treated first during the index procedure. Success is defined as ≤ 30% residual diameter stenosis without death or major complications.
* Absence of at least one patent native outflow artery.
* Presence of an aortic, iliac or femoral artificial graft.
* Failure to cross the target lesion with a guide wire. Successful crossing of the target lesion occurs when the tip of the guide wire is distal to the target lesion without the occurrence of flow-limiting dissection or perforation.
* Failure to successfully pre-dilate the target lesion. Successful pre-dilatation is defined as residual stenosis ≤ 70% with no flow-limiting dissection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Peak paclitaxel plasma concentration | Up to 30 days
  Paclitaxel plasma levels will be assessed at baseline, immediately post-index procedure, at 1h, 2h, 4h, 12h (or upon discharge), and 30 days post-index procedure.

SECONDARY OUTCOMES:
Area under the drug concentration time curve | Up to 30 days
  Area under the drug concentration time curve from the time of intervention to the time where the paclitaxel level is no longer quantifiable will be measured. Paclitaxel plasma levels will be assessed at baseline, immediately post-index procedure, at 1h, 2h, 4h, 12h(or upon discharge), and 30 days post-index procedure.
Technical success | At procedure
  Technical success, defined as successful delivery, inflation, deflation and retrieval of the intact study balloon device.
Device success | At procedure
  Device success, defined as achievement of < 50% residual stenosis of the target lesion (by core lab assessed quantitative angiography (QA)) using only the study device.
Procedure success | At procedure up to 12 hours
  Procedure success, defined as achievement of < 50% residual stenosis of the target lesion (by core lab assessed QA) using the study device with or without the use of additional devices, without the occurrence of death, amputation or repeat revascularization of the target vessel during index hospital stay.
Resting ankle brachial index | within 90 days of index procedure, and at 6, 12, 24 and 36 months post-index procedure
Change in Rutherford classification | baseline, 30 days, 6, 12, 24, and 36 months
Change in 6-minute walk test | baseline, 30 days, 6, 12, 24, and 36 months
Primary patency | 6 months
  defined as freedom from clinically-driven target lesion revascularization (TLR) and freedom from restenosis. Restenosis is defined by Duplex Ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥ 2.5 (core lab assessed) or by ≥ 50% stenosis by QA (core lab assessed)
Continuous DUS Peak systolic velocity ratio (PSVR) as measured by Duplex ultrasound | 30 days, 6, 12, 24, and 36 months
Late lumen loss | baseline, 6 months
  Defined as the difference in minimum luminal diameter of the target lesion between the index intervention and 6-month angiographic follow-up.
Quality of life | baseline, 30 days, 6, 12, 24, and 36 months
  Assessed by Change in walking Impairment Questionnaire (WIQ) scores
Evidence of Paclitaxel toxicity | At hospital discharge, 30 days
  Evidence of paclitaxel toxicity (rash, myelosuppression on blood counts, hepatitis, neuromuscular changes, hypotension, electrocardiogram (ECG) abnormalities, or gastrointestinal upset).
Major vascular complications | At hospital discharge, 30 days
Thrombolysis in Myocardial Infarction (TIMI)-defined major and minor bleeding | At hospital discharge, 30 days
Major adverse events | 30 days, 6, 12, 24, and 36 months
  defined as a composite of death, index limb amputation and TLR
All-cause death | 30 days, 6, 12, 24, and 36 months
Index limb above the ankle amputation | 30 days, 6, 12, 24, and 36 months
Index limb below the ankle amputation | 30 days, 6, 12, 24, and 36 months
Clinically-driven TLR | 30 days, 6, 12, 24, and 36 months
Clinically-driven target vessel revascularization (TVR) | 30 days, 6, 12, 24, and 36 months
Arterial thrombosis of the treated segment on angiography | 30 days, 6, 12, 24, and 36 months
Embolic events of the index limb | 30 days, 6, 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Metzger, MD, FACC, FSCAI, Principal Investigator — Wellmont CVA Heart Institute
Locations (3):
- United States (3):
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Wellmont Health System, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided